CLINICAL TRIAL: NCT03245112
Title: Retrospective Data Collection and Analysis of the Therapeutic Effect of Eribulin for Advanced Breast Cancer Patients.
Brief Title: Halaven Patient Registry (Metastatic Breast Cancer, MBC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Kaohsiung Breast Cancer Prevention and Education Society (KBCPES) (Unknown); Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 201700596B0
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Eribulin Mesylate — The patients received intravenous eribulin 1.4 mg/m2 over 2-5 minutes on days 1 and 8 of every 21 days.
  Other Names: Halaven

SUMMARY:
Since the first marketing authorization in the world in November 2010 granted by US FDA, Halaven has been approved for clinical use in more than 40 countries worldwide, including many Asian countries, e.g. Hong Kong, India, Japan, Malaysia, Myanmar, Philippines, South Korea, Singapore, Taiwan and Thailand. According to two large global phase III study reports of Halaven, very few Asian patients participated in these studies. In a phase II study of Halaven with metastatic breast cancer, the clinical efficacy and toxicity were reported only in 80 Japanese patients. Halaven has been granted its marketing authorization in Singapore since February 2011. However, most of other Asian countries including India have had the approval and launched from middle year of 2013 or in early 2014. Limited information of Halaven using in Asian patients are available except several case experience exchange presented by individual medical centers or as personal experience in the past. Some clinical concerns related to Halaven use are raised by clinicians during their clinical practice, such as how Halaven works on Asian patients, which type of patient obtains better clinical benefit from Halaven, and what are the main treatment related toxicities in Asian which may differ from Westerners due to potential ethnic diversity. Further understanding of Halaven related clinical benefit and toxicity in Asian patients through collecting clinical experience among Asian countries becomes necessary and may provide better information to anticipate these concerns.

The proposed "Halaven Patient Registry" (called the "Registry") will be a patient population-based registry to collect therapeutic related information from patients with metastatic breast cancer who were treated with Halaven that was given as a clinical decision by patient's treating physician based on clinical status of a patient and proper indication of Halaven and to gain a better understanding of the use of Halaven in such Asian patients.

ELIGIBILITY:
Inclusion Criteria:

* An eligible patient to be entered into the Registry is defined as:

  1. Patient with advanced breast cancer.
  2. Halaven was given or has been treating during the period of 1 Jan 2015 to 31 Dec 2016.
  3. Halaven was given as single or combination.
  4. Patient received at least one cycle treatment (a 21-day cycle or 2 doses) of Halaven.
  5. Patient with at least 80% of the required information of the Registry CRF to be entered. It will be calculated automatically by the Registry system.

     Patient to be selected for the Registry will be based on chorological order of a patient occurred in a study center during the defined period of the Registry, if all other eligibility criteria are met.

     Exclusion Criteria:
* Those who not meet the inclusion criteria will be excluded.

Ages: 24 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The advanced or metastatic breast cancer patient who received at least 1 course Halaven therapy was eligible to this study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-03-03 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 24 months
  he percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention

SECONDARY OUTCOMES:
Number of patients with adverse events | 24 months
  An AE may consist of the following: A new event which was not pre-existing at initial study drug administration. A pre-existing event which recurs with increased intensity or increased frequencysubsequent to study drug administration. An event which is present at the time of study drug administration which isexacerbated following initial study drug administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided